CLINICAL TRIAL: NCT01046045
Title: Impact and Efficacy of Everolimus Rescue Immunosuppression in the Treatment of Chronic Allograft Dysfunction in Renal Transplant Recipients
Brief Title: Everolimus Rescue Immunosuppression in the Treatment of Chronic Allograft Dysfunction in Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chow Kai Ming, Associate Consultant, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2008.004-T
Record Dates: First submitted 2010-01-06; First posted 2010-01-11 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Chronic Allograft Dysfunction in Renal Transplantation
Keywords: mammalian target-of-rapamycin inhibitors; chronic allograft dysfunction; everolimus; calcineurin inhibitors
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus (Active Comparator): before and after everolimus; in other words, comparison of specified outcome before and after treatment with everolimus
  Interventions: Drug: everolimus
- Calcineurin-inhibitor immunosuppression (Active Comparator): Cyclosporin-based immunosuppression without everolimus
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus — everolimus at an initial daily loading dose between 1 and 4 mg dose of everolimus will be adjusted to maintain a trough everolimus level between 5 and 12 ng/mL
  Other Names: Certican

SUMMARY:
Despite the remarkable improvement in short-term patient and graft survival among the recipients of kidney transplants, the progressive renal dysfunction (chronic allograft dysfunction) accompanied by chronic interstitial fibrosis, tubular atrophy, vascular occlusive changes and glomerulosclerosis remains the chief cause of graft loss. As a result of this damage from immunologic and non-immunologic injury, the long-term survival of kidney transplants has changed little during the past decade. And, among the non-immunologic factors, calcineurin inhibitor nephrotoxicity has been shown to be the most common factor leading to long-term graft damage and progression to graft failure. This is further supported by the previous finding that long-term use of calcineurin inhibitor-based therapy leads to deterioration in kidney function, even in recipients of non-renal organ transplants.

The growing interest in calcineurin inhibitor minimisation protocols to optimize renal transplant outcome offers a new therapeutic options in the management of patients with chronic allograft dysfunction. Recently, mammalian target-of-rapamycin inhibitors (mTOR inhibitors) including everolimus has been shown to achieve an improvement of long-term function through an early modulation of immunosuppressive regimen. In this aspect, percutaneous renal graft biopsy represents an important diagnostic tool to allow visualization of the lesions of chronic allograft dysfunction and therefore the ability to delineate the potential improvement after introduction of everolimus. Histologic and morphometric findings from a protocol-mandated biopsies obtained from renal transplant recipients who are suffering from chronic allograft dysfunction and treated with everolimus are needed to provide a clinical blueprint for the drug's efficacy, if confirmed.

DETAILED DESCRIPTION:
The objective of the present study is to evaluate the a priori hypothesis that calcineurin inhibitor and rescue immunosuppression with everolimus-based therapy would attenuate the renal parenchymal injury associated with long-term use of calcineurin inhibitors in renal transplant recipients with declining kidney function. Another objective of this study is to elucidate the efficacy of our approach to arrest the progression of allograft dysfunction by means of protocol renal allograft biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Biopsy-confirmed chronic allograft dysfunction or chronic allograft nephropathy, in the absence of acute rejection episode within the preceding 2 months
* Proteinuria < 0.8 g/day (or spot urine protein < 0.8 g/g-Cr) in 2 consecutive samples within 8 weeks
* Serum creatinine < 220 μmol/L or estimated glomerular filtration rate > 40 ml/min/1.73m2 by the Nankivell formula, which had been validated in kidney transplant recipients; this equation was expressed for use with a standard serum creatinine assay: glomerular filtration rate = 6.7/(standardized serum creatinine in μmol/L / 1000) + weight (kg)/4 - urea (mmol/L)/2 - 100 / height2 (m) + 35 if the subject is male (or 25 if the subject is female)
* Willingness to give written consent and comply with the study protocol

Exclusion Criteria:

* Pregnancy, lactating or childbearing potential without effective method of birth control
* Severe gastrointestinal disorders that interfere with their ability to receive or absorb oral medication
* Serum cholesterol > 7.8 mmol/L and/or serum triglycerides > 4.5 mmol/L despite lipid-lowering agents before conversion
* Systemic infection requiring therapy at study entry
* Participation in any previous trial on everolimus or sirolimus
* Patients receiving treatment of sirolimus or everolimus for other medical reasons within the past 12 months
* On other investigational drugs within last 30 days
* History of a psychological illness or condition such as to interfere with the patient's ability to understand the requirement of the study
* History of non-compliance
* Chronic lung disease
* Known history of sensitivity or allergy to everolimus

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-04; Primary Completion 2011-11 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
change in glomerular filtration rate decline rate and histological degree of fibrosis before and after treatment with everolimus | 12 months

SECONDARY OUTCOMES:
estimated glomerular filtration rate at 12 months | 12 months
morphometric studies | 12 months
cytokines before and after everolimus conversion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kai Ming Chow, MBChB, Principal Investigator — Chinese University of Hong Kong, Prince of Wales Hospital
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong